CLINICAL TRIAL: NCT02363257
Title: Compliance, Perceptions and Attitudes of Bus Employees and Commuters Towards Smoke Free Bus Policy (as Part of Smoke Free Public Places) in Mumbai, India
Brief Title: Smoke Free Policy Among BEST Bus Employees and Commuters in Mumbai
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Sharmila Pimple, Professor & Physician, Department of Preventive Oncology, Tata Memorial Hospital
Other Study IDs: 1369 BEST-SF
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Compliance
Keywords: Smoke free bus policy; BEST commuters; BEST employee
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Three years since the Smoke Free Mumbai campaign and six years since the ban on smoking in public places was implemented. It is necessary to review the situation at this point in time so that corrective actions if necessary can be taken. Hence, this study is planned to understand the perceptions and attitudes of commuters and bus employees (drivers, conductors and ticket checkers) regarding the law, its implementation, reactions from the commuters, violations observed, violations reported.

This study will help evaluate the implementation of provision of prohibiting smoking in public places and help understand how to increase the compliance. The results will inform enforcement and public health agencies about where to target enforcement and public education resources.

DETAILED DESCRIPTION:
Aim:-1.To assess the knowledge and awareness about tobacco legislation with specific reference to smoke free public places and understand the perceptions and attitude regarding implementation of smoke free BEST policy among BEST employees (mainly drivers, conductors and ticket checkers) in Mumbai. (in terms of reactions from commuters, violations observed, violations reported etc.).

2.Determine the Knowledge, attitudes and perception of BEST commuters about the provisions of smoke free public places and the smoke free public transport.

3.To identify the stakeholder challenges in implementation of the smoke free public transport system in Mumbai 4.To study the compliance with smoke free BEST policy by random observations at the BEST buses, depots and bus stops.

Study Design:

1. A cross sectional survey design to assess Knowledge, attitudes and perception about Section 4 of COTPA among BEST employees and BEST commuter
2. Observational design for assessment of compliance to smoke free public transport system (BEST) using a structured compliance tool.

Study Methodology:

1. Around 500 BEST employees, 500 BEST commuters and 25 management staff responsible for implementation check, in Mumbai will be enrolled after explaining the programme and obtaining informed consent. They will be interviewed by trained Social Workers using a validated structured questionnaire to collect information about their Knowledge and perceptions about provisions with in COTPA 2003 for Smoke free Public Places and perceived challenges with regards to implementation of smoke free public transport with specific reference to smoke free BEST buses.
2. Observation and reporting regarding compliance to smoke free public places using validated observational study tools will be conducted at 100 randomly selected BEST buses, 100 bus stops and all 26 bus depots.
3. Observational study tool will consist of the following observations for Compliance to Smoke free BEST Public Transport system.

   1. Presence of no smoking signage: Any pictorial, graphical or textual message displayed in a public place, which warns that smoking is prohibited in a public place, will be recorded as a signage.
   2. Compliance with specifications, as prescribed by COTPA for size, textual content, colour, font and design
   3. Absence of active smoking: At the time of observation.
   4. Absence of cigarettes butts or bidi ends: In Buses, Bus depots and Bus stops.

Definition of Public Places under BEST Bus transport system :

For the purpose of the surveys, the public places under BEST Bus transport system were grouped into three broad categories,

1.BEST Buses 2.BEST Bus Depots, office premises 3. BEST Bus Stops.

Stakeholders to be interviewed to know their views regarding challenges in implementation of the smoke free public transport system in Mumbai

1. BEST Committee members
2. Important people in the managerial and administrative cadre in authoritative positions who can influence tobacco policy
3. Members of Employee Unions within the organization
4. Medical Unit including - Chief Medical Officers, Junior and Senior Medical Officers, Paramedical workforce
5. BEST Commuters Forum
6. Personnel in authoritative positions in: G. M. office
7. Welfare Department
8. Personnel Department
9. PRO Department
10. Legal Department
11. BEST Commuters
12. Any other stakeholders eventually identified

Sampling Methodology:

The list of Bus Depots, Public transport Buses with routes and Bus stops will be prepared with the help of BEST undertaking. Category wise sample of 100 BEST buses, 100 bus stops and all 26 bus depots will be selected through a simple random sampling method .

Times of day for Compliance Survey data collection. There is no best prac¬tice for the time of day for observing compliance. One alternative is to visit venues at peak business hours to assess compliance when the most number of people are affected. Alternatively, venues could be visited at different times of the day.

The present study will collect data at three time sets viz: Morning 9.00- 11.00 am, Afternoon 2.00 -4.00 pm and Evening 5.00-7.00 pm to determine if compliance varies by time of day. The data collection tool will record the time of day of the visit.

Informed consent: Trained Medical Social Workers will administer the informed consent forms to the study participants in the presence of a witness Questionnaire administration Validated pre tested survey questionnaire will be administered to BEST employees and BEST commuters by trained Field investigators to record personal details, self tobacco consumption, knowledge about legislation for Smokefree Public places and perceived challenges in implementing the same.

Observation for Compliance:

Field investigators will be trained to observe violations and to record these on the designed format, for noting the compliance and violations at randomly selected BEST buses, bus stops and bus depots.

Outcome measures Analysis of Observational Data will measure the following outcomes.

1. The overall rate of compliance for all loca¬tions (Public place) visited.
2. The compliance rate for each category of location
3. Overall Compliance on each criteria / parameter selected for recording compliance as per protocol for all locations.
4. The compliance rate for each criteria / parameter selected for recording compliance for each category of location.

Statistical Analysis Data entry will be done in the Department of Preventive Oncology, Tata Memorial Hospital using SPSS version 18. High quality data collection will be ensured with regular checks for data collection and data entry for completeness and consistency across responses. Descriptive statistics will be used to record compliance, perceptions and attitudes regarding implementation of smoke free BEST policy. Both descriptive and inferential statistics will be generated for describing variables under the study objectives. Interview data will be qualitative in nature and will be analyzed to determine themes from respondents and to identify variations in responses to questions about smoke-free compliance issues. Multivariate analysis will be performed to identify the factors determining compliance to the law .

Benefits:

This project will increase awareness of the BEST employees regarding the law. Results of the study will inform policymakers how well the law is being complied with and the link between the levels of compliance found and resources needed to im¬prove or maintain compliance with smoke-free public places.

Outcomes of the study will help enforcement agencies to take up result oriented measures and also to create greater pressure for action for effective enforcement.

Study will provide information to Managers of the locations visited about overall compli-ance and can be used to design compliance checks that can be conducted at regular intervals and encourage them to comply with the law.

Study results can inform General public/ commuters about lev¬els of compliance with the law, encourage the public to comply with the law, and call for ongoing or increased enforcement of the law by the government.

Proper implementation of the law will help in reducing exposure to second hand smoke, reducing the environmental impact of unsightly litter such as cigarette butts and packets and providing supportive environments for non-smokers and for those attempting to quit smoking. Creating smoke-free outdoor areas, such as public transport stops and stations, can support those who have quit and make smoking less visible to children and young people.

ELIGIBILITY:
Inclusion Criteria:

* BEST employees (Bus drivers, Bus conductors and ticket checkers) and regular BEST commuters (>18 years) in Mumbai will be invited to participate in the study.

Exclusion Criteria:

* BEST employees and Commuters refusing to participate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BEST Employees, Regular BEST commuters, Stakeholders:1.BEST Committee members 2.Important people in the managerial and administrative cadre in authoritative positions who can influence tobacco policy 3.Members of Employee Unions within the organization 4.Medical Unit including - Chief Medical Officers, Junior and Senior Medical Officers, Paramedical workforce 5.BEST Commuters Forum 6.Personnel in authoritative positions in: G. M. office 7.Welfare Department 8.Personnel Department 9.PRO Department 10.Legal Department 11.BEST Commuters 12.Any other stakeholders eventually identified
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Compliance and Interview | 2 years
  The overall rate of compliance for all locations (Public place) visited.
  3.
Compliance and Interview | 2 years
  The compliance rate for each category of location
Compliance and Interview | 2 years
  Overall Compliance on each criteria / parameter selected for recording compliance as per protocol for all locations.
Compliance and Interview | 2 years
  The compliance rate for each criteria / parameter selected for recording compliance for each category of location.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sharmila A Pimple, MD, Principal Investigator — Tata Memorial Centre